CLINICAL TRIAL: NCT04045821
Title: Endometrial Response Following Use of the Stem Cell Mobilizing Agent AMD3100 in a Population of Infertile Women With a Thin Endometrial Lining
Brief Title: Endometrial Rejuvenation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMA-2019-02
Record Dates: First submitted 2019-07-25; First posted 2019-08-06 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Infertility of Uterine Origin
MeSH Terms: interventions — plerixafor; Saline Solution; Dilatation and Curettage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Patients in this arm will not receive the study drug. A placebo of normal saline will be injected subcutaneously and the D&C procedure will be completed.
  Interventions: Drug: Normal saline; Procedure: dilation and curettage
- Intervention (Experimental): Patients in this arm will receive a dose of the study drug, AMD3100, injected subcutaneously and the D&C procedure will be completed.
  Interventions: Drug: AMD3100; Procedure: dilation and curettage

INTERVENTIONS:
Drug: AMD3100 — Subjects in this arm will have AMD3100 administered per the standard dosing regimen of 0.24 mg/kg actual body weight subcutaneous x1 dose
  Arms: Intervention
Drug: Normal saline — Subjects in this arm will have a placebo of normal saline administered subcutaneously x1 dose
  Arms: Control
Procedure: dilation and curettage — all participants will undergo routine D&C procedure
  Other Names: D&C

SUMMARY:
To evaluate the response of the endometrial lining after subcutaneous administration of the medication AMD3100. This medication mobilizes stem cells and will be used in a population of infertile women with a thin endometrium who are undergoing frozen-thawed embryo transfer. The investigators will assess associations between response to stem cell mobilization and pregnancy outcomes.

DETAILED DESCRIPTION:
This study seeks to help each participant build a better endometrial lining which is suitable to implantation and maintenance of a healthy pregnancy. While animal models demonstrating the effectiveness of stem cell recruitment on improved endometrial thickness and pregnancy outcomes are plentiful, human studies are lacking. The use of stem cells from the peripheral circulation in humans could potentially allow for enhanced endometrial proliferation. The objective of this study is to perform a prospective randomized, controlled trial to evaluate the response of the endometrial lining after subcutaneous administration of AMD3100 (plerixafor). AMD3100 is an immunostimulant used to mobilize hematopoietic stem cells in the bloodstream. This intervention will be studied in a population of infertile women with a thin endometrium who have failed previous embryo transfer cycles and are undergoing a frozen-thawed embryo transfer. This study seeks to evaluate both the endometrial response to stem cell mobilization via AMD3100 as well as pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients planning to undergo a frozen-thawed embryo transfer cycle using a single euploid blastocyst.
2. Patients who have previously undergone at least 2 unsuccessful frozen-thawed embryo transfer cycles, defined as failure to achieve a clinical pregnancy (visualization of intrauterine gestational sac on ultrasound) or a cancelled embryo transfer cycle due to inadequate endometrial thickness.
3. Patients with a diagnosis of thin endometrial lining (less than 6 mm maximum thickness) during at least one prior unsuccessful embryo transfer cycle.
4. Initiation of the most recent unsuccessful frozen-thawed embryo transfer cycle with a thin endometrial lining must have occurred after January 1, 2017.

Exclusion Criteria:

1. Fewer than 2 prior unsuccessful frozen-thawed embryo transfer cycles.
2. Most recent unsuccessful frozen-thawed embryo transfer prior to January 1, 2017.
3. No euploid embryos available for transfer.
4. Mullerian anomalies, excluding arcuate uterus
5. Submucosal fibroids
6. History of uterine surgery, excluding polypectomy, D&C, and Cesarean section
7. Communicating hydrosalpinx without plans for surgical correction prior to study enrollment.
8. Failure of patient to agree to enrollment in study with written consent.
9. History of drug sensitivity or adverse reaction to AMD3100 (plerixafor).
10. Pregnancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all participants must be biologically female and possess a uterus
Enrollment: 3 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness | measured on day prior to progesterone initiation during frozen embryo transfer cycle
  measurement of endometrial thickness

SECONDARY OUTCOMES:
number of participants with a chemical pregnancy | 9-11 days post embryo transfer
  defined by a positive bHCG
number of participants with a clinical pregnancy | seen as early as 18 days post embryo transfer
  defined as the presence of an intrauterine gestational sac
number of participants with a live births | typically 9 months from embryo transfer
  number of deliveries resulting from embryo transfer
endometrial volume | measured at baseline visit during cycle 1 (one month) and after progesterone initiation during cycle 4 (one month)
  measurement of uterine endometrium based on 3D ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Brent Hanson, MD, Study Director — Reproductive Medicine Associates of New Jersey
Locations (3):
- United States (3):
  - Reproductive Medicine Associates of Northern California, San Francisco, California
  - Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey
  - Reproductive Medicine Associates of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No